CLINICAL TRIAL: NCT02973074
Title: Pilot Study for Investigation of the Feasibility and for Optimization of Oral Iron Substitution in the Course of Patient Blood Management for Orthopedic Surgery
Brief Title: Oral Iron Substitution for Orthopedic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no enough partícipants enrolled in the 1 year planned for recruitment
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Nina Pauker, MD, Dr. med. univ., Kepler University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-124-16
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency; patient blood management; anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OLEOvital (Other): 30mg iron are being administered orally twice a day for a period of 4 Weeks it is a granulated powder which is taken orally and then solved with saliva, without taking water
  Interventions: Dietary Supplement: OLEOvital

INTERVENTIONS:
Dietary Supplement: OLEOvital — 2sachets with 30mg iron per day for a 4 weeks period

SUMMARY:
The aim of this pilot study is to investigate an 4 weeks period of oral iron substitution in the course of Patient Blood Management in preparation for orthopedic surgery.

DETAILED DESCRIPTION:
Patient blood management (PBM) is a clinical multidisciplinary, patient orientated concept for treatment of anaemia, reduction of intraoperative blood loss and increasing anaemic tolerance.

In the Kepler University Hospital (former General Hospital Linz) PBM was introduced in 2006. Since then patients for elective orthopedic surgery (knee an hip replacement) are screened for iron deficiency anaemia and if needed treated with the more effective intravenous iron.

Oral iron medications are not as efficient (low bioavailability, more side effects) as the intravenous iron infusion. Although there is risk of anaphylactoid reactions.

In this study the new oral iron supplement OLEOvital Eisen forte (available in Austria) ist tested on its effectivity for treatment of iron deficiency in the course of PBM.

It has a much more higher bioavailability without the typically side effects of the routinely used oral iron medications.

Within this study the investigators want to examine the feasibility of this iron substitution concept OLEOvital and its efficacy. Also the investigators want to get pilot data for a further randomized controlled trial.

The increase of the hemoglobin level in 4 weeks of minimum 1g/dl is going to be expected and monitored.

For comparison of the new oral substitution concept OLEOvital with the standard intravenous iron substitution an historic control group is going to be used.

ELIGIBILITY:
Inclusion Criteria:

* age over 55 years
* indication for patient blood management for elective orthopedic surgery
* listed for a orthopedic surgery (e.g. hip or knee replacement) 5-7 weeks after begin of patient blood management
* Haemoglobin male < 12-13g/dl, female <11-12g/dl
* written informed consent after written and verbal information

Exclusion Criteria:

* indication for treatment with erythropoietin
* pregnancy
* nursing period
* diarrhea or tendency to diarrhea
* fructose intolerance
* pre - menopause
* permanent or expected blood loss
* participation in other study
* expected compliance problems
* legal incapacity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-25; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
increase of hemoglobin level | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Meier, Prof. Dr., Principal Investigator — Kepler University Hospital Linz, Clinic for Anesthesiology and intensive care medicine
Locations (1):
- Kepler University Hospital, Linz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gombotz H, Rehak PH, Shander A, Hofmann A. Blood use in elective surgery: the Austrian benchmark study. Transfusion. 2007 Aug;47(8):1468-80. doi: 10.1111/j.1537-2995.2007.01286.x. PMID 17655591
- [Background] Seicean A, Alan N, Seicean S, Neuhauser D, Weil RJ. The effect of blood transfusion on short-term, perioperative outcomes in elective spine surgery. J Clin Neurosci. 2014 Sep;21(9):1579-85. doi: 10.1016/j.jocn.2014.03.003. Epub 2014 May 19. PMID 24852902
- [Background] Danninger T, Rasul R, Poeran J, Stundner O, Mazumdar M, Fleischut PM, Poultsides L, Memtsoudis SG. Blood transfusions in total hip and knee arthroplasty: an analysis of outcomes. ScientificWorldJournal. 2014 Jan 21;2014:623460. doi: 10.1155/2014/623460. eCollection 2014. PMID 24587736
- [Background] Meybohm P, Richards T, Isbister J, Hofmann A, Shander A, Goodnough LT, Munoz M, Gombotz H, Weber CF, Choorapoikayil S, Spahn DR, Zacharowski K. Patient Blood Management Bundles to Facilitate Implementation. Transfus Med Rev. 2017 Jan;31(1):62-71. doi: 10.1016/j.tmrv.2016.05.012. Epub 2016 May 28. PMID 27317382